CLINICAL TRIAL: NCT05928182
Title: El Faro: Addressing Mental Health Inequities Among Latinx Children With ADHD in Durham
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00111427
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2023-11

CONDITIONS: ADHD; Psychiatric Health
Keywords: Psychiatric Health; Children; ADHD; Latinx Community
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: All participants will receive treatment and symptom severity will be measured pre and post-treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Participants (Experimental): Active treatment group participants
  Interventions: Behavioral: El Faro Treatment Intervention

INTERVENTIONS:
Behavioral: El Faro Treatment Intervention — Pre - Measures: complete Child Behavior Checklist (CBCL), ADHD module of the MINI International Neuropsychiatric Interview for Children and Adolescents (MINI) administered by study team, ADHD Rating Scale (ADHD-RS; parent and teacher ratings), ADHD Functional Impartment Scale (ADHD-FX), Parenting Sense of Competence (PSOC), demographic information, and medical history. [All rating scales are parent-report unless noted otherwise]
  Treatment: Complete an 8-week adapted El Faro treatment intervention with homework tasks.
  Post-Measures: CBCL, ADHD-RS (parent and teacher ratings), ADHD-FX, and PSOC. We will also acceptability and feasibility via measuring session attendance (rated by the therapist each session), homework completion (rated by the therapist each session), 7 treatment acceptability questions. [All rating scales are parent-report unless noted otherwise and administered at post-treatment visit unless noted otherwise].

SUMMARY:
Study team members from El Futuro in Durham, North Carolina have created an intervention called El Faro. El Faro helps Latinx families of children with ADHD understand and cope with the stress and difficulties presented by the disorder. We propose to develop a community-engaged research partnership between El Futuro and the Duke ADHD Program that aims to pilot-test an adapted El Faro treatment.

ELIGIBILITY:
Inclusion Criteria:

* Child is between the ages of 6 to 12 years
* Child has received a previous diagnosis of ADHD in the community based on caregiver report
* ADHD Rating Scale (parent rating scale of ADHD symptoms) symptom severity score of 24 or higher
* Child meets DSM-5 criteria for ADHD (any presentation) based on the MINI
* Generally healthy (i.e., no major medical problems that will interfere with study participation)
* Caregiver's willingness to keep any current psychiatric medication regimen for child diagnosed with ADHD constant throughout the study duration
* Caregiver age 18 years and older
* Caregiver self-identify as Latinx

Exclusion Criteria:

* Caregiver's child has previous diagnosis of Autism, Schizophrenia, or Bipolar Disorder in the community per caregiver report or other psychiatric disorder that is primary to ADHD or may interfere with study involvement.
* Caregiver unable to attend all El Faro sessions
* Plan to initiate new ADHD treatment for identified child with ADHD during study participation (previously established ADHD treatments are allowable)
* Other concerns besides ADHD that would interfere with study participation according to the study team.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Preliminary Treatment Efficacy of adapted EL Faro as measured by change in the ADHD Rating Scale (ADHD-RS) | (8 weeks)
  An 18-item questionnaire with a 4-point Likert scale ranging from Never or Rarely (0) - Very Often (3). With a total score range of 0 -54. A lower score indicated a better outcome.
Preliminary Treatment Efficacy of adapted EL Faro as measured by change in the ADHD Functional Impairment Scale (ADHD-FX) | (8 weeks)
  A 32-item questionnaire with 4-point Likert scale ranging from Not at All (0) - A lot (3). With a total score range of 0 - 96. A lower score indicates better outcome.
Preliminary Treatment Efficacy of adapted EL Faro as measured by change in the Attention Problem Scale of the Child Behavior Checklist (CBCL) | (8 weeks)
  A 10-item parent report questionnaire with a 3-point Likert Scale ranging from Not True (0) to Very True or Often True (2). A total score range of 0-20. Lower scores indicate better outcomes.
Preliminary Treatment Efficacy of adapted EL Faro as measured by change in the ADHD Scale of the Child Behavior Checklist (CBCL) | (8 weeks)
  A 7-item parent report questionnaire with a 3-point Likert Scale ranging from Not True (0) to Very True or Often True (2). A total score range of 0-14. Lower scores indicate a better outcome.
Preliminary Treatment Efficacy of adapted EL Faro as measured by change in the Parenting Sense of Competence Scale (PSOC) | (8 weeks)
  A 16-item questionnaire with a 6-point Likert scale ranging from Strongly Disagree (1) - Strongly Agree (6). A total score range of 16 - 96. A higher score indicates a better outcome.
Feasibility of adapted El Faro Treatment as measured by percentage of attrition | (8 weeks)
  Attrition of <25% will be set to establish feasibility
Feasibility of adapted El Faro Treatment as measured by homework compliance | 8 weeks
Acceptability of adapted El Faro Treatment as measured by how satisfactory participants felt that the treatment was overall | 8 weeks
  Acceptability will be based on how satisfactory participants felt that the treatment was overall (ranging from 1-7 with 7 indicating the highest rating of treatment satisfaction)
Acceptability of adapted El Faro Treatment as measured by caregiver perceptions | 8 weeks
  Caregiver perceptions about the extent of ADHD psychoeducation they received, how the content was relevant to their experiences, whether the techniques introduced were understandable, if they were confident about regularly using the techniques taught, and if they would recommend El Faro to other families of children with ADHD (on a scale ranging from 1 = not at all to 4 = extremely).

CONTACTS AND LOCATIONS:
Overall Officials: John Mitchell, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no IPD for this study.

DOCUMENTS (1):
  • Informed Consent Form (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT05928182/ICF_000.pdf